CLINICAL TRIAL: NCT02177019
Title: Assessment of a Personalized Health Care Intervention for Frequent Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00050263; 1K18HS022443-01 (AHRQ)
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-05

CONDITIONS: Frequent Headaches
Keywords: frequent headaches; personalized health plan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Development of personal health plan (Experimental): Personal Health Plan
  Interventions: Other: Personalized health plan

INTERVENTIONS:
Other: Personalized health plan

SUMMARY:
The research project is a component of a mentored research career enhancement award. The purpose of the award is to help the PI and his collaborators prepare for future research grant opportunities through the Patient Centered Outcomes Research Institute (PCORI). The research project is a feasibility study with the following specific aims; 1) to assess outcomes associated with a personalized health plan for frequent headaches; 2) to identify measurable outcomes that are meaningful to patients with frequent headaches; and 3) to create a patient stakeholder group to inform patient-centered outcomes research for frequent headaches. Specific Aim #1 will be achieved by recruiting and enrolling 40 established patients at the Duke Family Medicine Center who have frequent headaches. The intervention consists of 3 study visits with the PI, 2 clinical consultations with subjects' established primary care provider at the Duke Pickens Family Medicine Center, and participation in 2 focus groups. Personalized health plans might consist of a combination of medical management, lifestyle changes, nutrition counseling, or other therapeutic modalities as appropriate. Data analysis will be descriptive; no formal hypotheses will be tested.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic headache

Exclusion Criteria:

* patients who do not understand english language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Daily headache scores, | Daily from baseline to 3 months
  Subjects will report daily headache scores to the CRC.
Change in Quality of life | Baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Remy Coeytaux, MD, Principal Investigator — Duke